CLINICAL TRIAL: NCT02255097
Title: A Phase II Clinical Trial of Single Agent Pembrolizumab (MK-3475) in Subjects With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC) Who Have Failed Platinum and Cetuximab
Brief Title: Study of MK-3475 (Pembrolizumab) in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma After Treatment With Platinum-based and Cetuximab Therapy (MK-3475-055/KEYNOTE-055)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-055; 2014-002447-18 (EudraCT Number)
Record Dates: First submitted 2014-09-30; First posted 2014-10-02 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for up to 24 months
  Interventions: Biological: pembrolizumab

INTERVENTIONS:
Biological: pembrolizumab
  Other Names: MK-3475; KEYTRUDA®

SUMMARY:
This is a study of single-agent pembrolizumab (MK-3475) in participants with recurrent and/or metastatic head and neck squamous cell carcinoma (HNSCC) who have progressed on platinum-based and cetuximab therapy. The primary study hypothesis is that pembrolizumab will provide a clinically meaningful objective response rate (ORR).

With protocol amendment 05 (02-Jan-2018), once study participants have achieved the study objective or the study has ended, participants will be discontinued from this study and enrolled in an extension study to continue protocol-defined assessments and treatment.

ELIGIBILITY:
Inclusion criteria:

* Histologically- or cytologically-confirmed recurrent or metastatic HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx that is considered incurable by local therapies
* Tumor progression or recurrence within 6 months of the last dose of any number of platinum-based and cetuximab therapy lines in the adjuvant, primary, recurrent, or metastatic setting; must be resistant (not responding) to both platinum and cetuximab
* Available tissue for biomarker analysis
* Measurable disease based on RECIST 1.1 as determined by central review
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function
* Female participants of childbearing potential must have a negative urine or serum pregnancy test and must be willing to use 2 adequate methods of contraception starting with the screening visit through 120 days after the last dose of pembrolizumab
* Male participants with a female partner(s) of childbearing potential must be willing to use 2 adequate methods of contraception from screening through 120 days after the last dose of pembrolizumab

Exclusion criteria:

* Disease that is suitable for local therapy administered with curative intent
* Currently receiving treatment in a study of an investigational agent or using an investigational device <= 4 weeks prior to the first dose of trial medication
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial medication
* Not recovered from AEs due to a previously administered therapy
* Known additional malignancy that is progressing or requires active treatment excluding basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Active, non-infectious pneumonitis
* Active infection requiring systemic therapy
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial medication
* Human immunodeficiency virus (HIV)
* Hepatitis B or C
* Received live vaccine within 30 days of planned start of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2014-10-24 (Actual); Primary Completion 2016-04-22 (Actual); Study Completion 2021-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Bauml J, Seiwert TY, Pfister DG, Worden F, Liu SV, Gilbert J, Saba NF, Weiss J, Wirth L, Sukari A, Kang H, Gibson MK, Massarelli E, Powell S, Meister A, Shu X, Cheng JD, Haddad R. Pembrolizumab for Platinum- and Cetuximab-Refractory Head and Neck Cancer: Results From a Single-Arm, Phase II Study. J Clin Oncol. 2017 May 10;35(14):1542-1549. doi: 10.1200/JCO.2016.70.1524. Epub 2017 Mar 22. PMID 28328302
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Guo T, Califano JA. Molecular biology and immunology of head and neck cancer. Surg Oncol Clin N Am. 2015 Jul;24(3):397-407. doi: 10.1016/j.soc.2015.03.002. Epub 2015 Apr 20. PMID 25979390
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were eligible to receive second course treatment with pembrolizumab if they met criteria for re-treatment. Per protocol, response or progression during the second course of pembrolizumab was not counted towards efficacy outcome measures and adverse events during the second course of pembrolizumab were not counted towards safety outcome measures.
Pre-assignment Details: Final analyses for all primary outcome measures were done at the protocol-specified primary outcome measure met date. The analyses for all secondary outcome measures and the collection of adverse events were updated at the end of study date.
  One participant allocated to receive pembrolizumab did not receive treatment. This participant was not eligible for safety or efficacy analysis.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 24 months. Participants who stopped pembrolizumab as a result of obtaining a confirmed complete response (CR) or those who stopped after receiving pembrolizumab for 24 months for reasons other than disease progression or intolerability, were eligible for up to an additional 1 year of treatment after progressive disease if they met the criteria for re-treatment.
Period: Overall Study
Arm/Group | Pembrolizumab
Started | 172
Treated | 171
Received Second Course of Pembrolizumab | 3
Completed | 0
Not Completed | 172
Not completed — Death | 151
Not completed — Lost to Follow-up | 5
Not completed — Participation in Study Discontinued by Sponsor | 8
Not completed — Withdrawal by Subject | 7
Not completed — Allocated but not treated | 1

BASELINE CHARACTERISTICS:
Population: The baseline population included all participants allocated to receive ≥1 dose of pembrolizumab.
Groups:
- Pembrolizumab: Participants received pembrolizumab 200 mg by IV infusion on Day 1 of each 3-week cycle for up to 24 months. Participants who stopped pembrolizumab as a result of obtaining a CR or those who stopped after receiving pembrolizumab for 24 months for reasons other than disease progression or intolerability, were eligible for up to an additional 1 year of treatment after progressive disease if they met the criteria for re-treatment.
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 153
  More than one race | 0
  Unknown or Not Reported | 0
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression status by immunohistochemistry assay using tumor tissue from an archival or newly obtained biopsy. Participants with a tumor proportion score (TPS) were classified as follows: ≥50% = PD-L1 strongly positive; 1-49% = PD-L1 weakly positive; and <1% = PD-L1 negative.
  Participants
    ≥50% | 44
    ≥1 - <50% | 77
    <1% | 46
    Unknown | 5

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: ORR was assessed by RECIST 1.1 by performing imaging every 6-9 weeks after the first dose of treatment. ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR) defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or Partial Response (PR) defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference. Participants with missing data were considered non-responders.
Time Frame: Up to 36 months
Population: All participants who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 171
Percentage of participants | 16.4 [11.2 to 22.8]
Statistical Analysis 1: Comparison: Pembrolizumab; Analysis comparing the ORR for pembrolizumab to a fixed efficacy target of 5% using an exact test of binomial distribution; Test type: Superiority or Other; p < 0.001, exact binomial distribution; null hypothesis (H0): p ≤ 0.05 versus alternate hypothesis (H1): p > 0.05

2. Primary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Strong Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a strong PD-L1 expression status were evaluated for ORR by RECIST 1.1. The expression of PD-L1 was determined by immunohistochemistry (IHC) and strong PD-L1 positive was defined as a PD-L1 tumor proportion score ≥50%. ORR was assessed by performing imaging every 6-9 weeks after the first dose of treatment. ORR was defined as the percentage of participants in the analysis population who had a CR defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or PR defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference. Participants with missing data were considered non-responders.
Time Frame: Up to 36 months
Population: All participants who received at least one dose of study treatment with a tumor proportion score ≥50%
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 44
Percentage of participants | 27.3 [15.0 to 42.8]
Statistical Analysis 1: Comparison: Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, exact binomial distribution; H0: p ≤ 0.05 versus H1: p > 0.05

3. Primary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of the product, whether or not considered related to the product. Worsening of a preexisting condition temporally associated with the use of the product was also an AE. A serious adverse event (SAE) was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, or was another important medical event. Per protocol, analysis for this outcome measure was planned to be performed during the initial (first) course of therapy only.
Time Frame: Up to 27 months
Population: All participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 171
Participants | 166

4. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an AE
Description: as for outcome 3
Time Frame: Up to 24 months
Population: All participants who received at least one dose of study treatment
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 171
Participants | 24

5. Secondary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a positive PD-L1 expression status were evaluated for ORR by RECIST 1.1. PD-L1 expression was determined by IHC and PD-L1 positive was defined as a PD-L1 tumor proportion score ≥1%. ORR was assessed by performing imaging every 6-9 weeks after the first dose of treatment. ORR was defined as the percentage of participants in the analysis population who had a CR defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or PR defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference. Participants with missing data were considered non-responders.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a tumor proportion score ≥1%
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 121
Percentage of participants | 18.2 [11.8 to 26.2]
Statistical Analysis 1: Comparison: Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, exact binomial distribution; H0: p ≤ 0.05 versus H1: p > 0.05

6. Secondary Outcome: Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Human Papillomavirus (HPV) Positive Tumors
Description: Participants with a HPV-positive tumor biopsy were evaluated for ORR by RECIST 1.1. ORR was assessed by performing imaging every 6-9 weeks after the first dose of treatment. ORR was defined as the percentage of participants in the analysis population who had a CR defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or PR defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference. Participants with missing data were considered non-responders.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a HPV-positive tumor
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 71
Percentage of participants | 14.1 [7.0 to 24.4]
Statistical Analysis 1: Comparison: Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0027, exact binomial distribution; H0: p ≤ 0.05 versus H1: p > 0.05

7. Secondary Outcome: Objective Response Rate (ORR) by Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: ORR was assessed by modified RECIST 1.1 by performing imaging every 6-9 weeks after the first dose of treatment. ORR was defined as the percentage of participants in the analysis population who had a CR defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or PR defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference. If imaging shows disease progression (PD) imaging was repeated 4 weeks later to confirm progression. PD was defined as at least a 20% increase in the sum of diameters of target lesions and new measurable lesions, taking as reference the smallest sum recorded since treatment started. Participants with missing data were considered non-responders.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 171
Percentage of participants | 16.4 [11.2 to 22.8]
Statistical Analysis 1: Comparison: Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, exact binomial distribution; H0: p ≤ 0.05 versus H1: p > 0.05

8. Secondary Outcome: Objective Response Rate (ORR) by Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a positive PD-L1 expression status were evaluated for ORR by modified RECIST 1.1. PD-L1 expression was determined by IHC and PD-L1 positive was defined as a tumor proportion score ≥1%. ORR was assessed by performing imaging every 6-9 weeks after the first dose of treatment. ORR was defined as the percentage of participants in the analysis population who had a CR defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or PR defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference. If imaging shows disease progression (PD) imaging was repeated 4 weeks later to confirm progression. PD was defined as at least a 20% increase in the sum of diameters of target lesions and new measurable lesions, taking as reference the smallest sum recorded since treatment started. Participants with missing data were considered non-responders.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a tumor proportion score ≥1%
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 121
Percentage of participants | 18.2 [11.8 to 26.2]
Statistical Analysis 1: Comparison: Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, exact binomial distribution; H0: p ≤ 0.05 versus H1: p > 0.05

9. Secondary Outcome: Objective Response Rate (ORR) by Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Strong Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a strong positive PD-L1 expression status were evaluated for ORR by modified RECIST 1.1. PD-L1 expression was determined by IHC and strong PD-L1 positive was defined as a tumor proportion score ≥50%. ORR was defined as the percentage of participants in the analysis population who had a CR defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm or PR defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference. If imaging shows disease progression (PD) imaging was repeated 4 weeks later to confirm progression. PD was defined as at least a 20% increase in the sum of diameters of target lesions and new measurable lesions, taking as reference the smallest sum recorded since treatment started. Participants with missing data were considered non-responders.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a tumor proportion score ≥50%
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 44
Percentage of participants | 27.3 [15.0 to 42.8]
Statistical Analysis 1: Comparison: Pembrolizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, exact binomial distribution; H0: p ≤ 0.05 versus H1: p > 0.05

10. Secondary Outcome: Response Duration (DOR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: DOR was based on RECIST 1.1 and measured from the time measurement criteria were first met for CR/PR (whichever was first recorded) until the first date that recurrent or PD was objectively documented (taking as reference for PD the smallest measurements recorded on study). DOR was censored at the last tumor assessment date if a responder did not have PD or death. Non-responders were not included in the analysis. The lower and upper limits were estimated at the time of data cutoff. DOR was analyzed by the Kaplan-Meier method for censored data and reported in months.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a best overall response as confirmed complete response or partial response
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 28
Months | 15.7 [2.8 to NA] — NA=Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

11. Secondary Outcome: Response Duration (DOR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a positive PD-L1 expression status were evaluated for DOR based on RECIST 1.1. PD-L1 expression was determined by IHC and PD-L1 positive was defined as a PD-L1 combined positive score ≥1%. DOR was measured from the time measurement criteria were first met for CR/PR (whichever was first recorded) until the first date that recurrent or PD was objectively documented (taking as reference for PD the smallest measurements recorded on study). DOR was censored at the last tumor assessment date if a responder did not have PD or death. Non-responders were not included in the analysis. The lower and upper limits were estimated at the time of data cutoff. DOR was analyzed by the Kaplan-Meier method for censored data and reported in months.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a combined positive score ≥1% and a best overall response as confirmed complete response or partial response
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 25
Months | 15.7 [2.8 to NA] — NA=Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

12. Secondary Outcome: Response Duration (DOR) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Strong Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a strong PD-L1 expression status were evaluated for DOR based n RECIST 1.1. PD-L1 expression was determined by IHC and strong PD-L1 positive was defined as a PD-L1 tumor proportion score ≥50%. DOR was measured from the time measurement criteria were first met for CR/PR (whichever was first recorded) until the first date that recurrent or PD was objectively documented (taking as reference for PD the smallest measurements recorded on study). DOR was censored at the last tumor assessment date if a responder did not have PD or death. Non-responders were not included in the analysis. The lower and upper limits were estimated at the time of data cutoff. DOR was analyzed by the Kaplan-Meier method for censored data and reported in months.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a tumor proportion score ≥50% and a best overall response as confirmed complete response or partial response
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 12
Months | 22.8 [4.2 to NA] — NA = Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse

13. Secondary Outcome: Progression-free Survival (PFS) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in All Participants
Description: PFS was defined as the time from the first day of study treatment to the first documented PD per RECIST 1.1 or death due to any cause, whichever occurred first. Using RECIST 1.1, PD was defined as either a 20% relative increase in the sum of diameters of target lesions, taking as reference the smallest sum on study OR an absolute increase of >5 mm the sum of lesions, OR the appearance of new lesions. PFS was analyzed by the Kaplan-Meier method for censored data and reported in months. Participant data were censored at last assessment.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 171
Months | 2.1 [2.1 to 2.1]

14. Secondary Outcome: Progression-free Survival (PFS) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a positive PD-L1 expression status were evaluated for PFS. PD-L1 expression was determined by IHC and PD-L1 positive was defined as a PD-L1 combined positive score ≥1%. PFS was defined as the time from the first day of study treatment to the first documented PD per RECIST 1.1 or death due to any cause, whichever occurred first. Using RECIST 1.1, PD was defined as either a 20% relative increase in the sum of diameters of target lesions, taking as reference the smallest sum on study OR an absolute increase of >5 mm the sum of lesions, OR the appearance of new lesions. PFS was analyzed by the Kaplan-Meier method for censored data and reported in months. Participant data were censored at last assessment.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a combined positive score ≥1%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 141
Months | 2.1 [2.0 to 2.1]

15. Secondary Outcome: Progression-free Survival (PFS) by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) in Strong Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a strong PD-L1 expression status were evaluated for PFS by modified RECIST 1.1. PD-L1 expression was determined by IHC and strong PD-L1 positive was defined as a PD-L1 tumor proportion score ≥50%. PFS was defined as the time from the first day of study treatment to the first documented PD per RECIST 1.1 or death due to any cause, whichever occurred first. Using RECIST 1.1, PD was defined as either a 20% relative increase in the sum of diameters of target lesions, taking as reference the smallest sum on study OR an absolute increase of >5 mm the sum of lesions, OR the appearance of new lesions. PFS was analyzed by the Kaplan-Meier method for censored data and reported in months. Participant data were censored at last assessment.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a tumor proportion score ≥50%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 44
Months | 2.1 [1.8 to 3.6]

16. Secondary Outcome: Overall Survival (OS) in All Participants
Description: OS was defined as the time from the first day of study treatment to death due to any cause. OS was analyzed by the Kaplan-Meier method for censored data and reported in months. Participant data were censored at last assessment.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 171
Months | 8.5 [6.6 to 11.1]

17. Secondary Outcome: Overall Survival (OS) in Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a positive PD-L1 expression status were evaluated for OS. PD-L1 expression was determined by IHC and PD-L1 positive was defined as a PD-L1 combined positive score ≥1%. OS was defined as the time from the first day of study treatment to death due to any cause. OS was analyzed by the Kaplan-Meier method for censored data and reported in months. Participant data were censored at last assessment.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a combined positive score ≥1%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 141
Months | 9.0 [6.2 to 11.8]

18. Secondary Outcome: Overall Survival (OS) in Strong Programmed Cell Death Ligand 1 (PD-L1) Positive Participants
Description: Participants with a strong PD-L1 expression status were evaluated for OS. PD-L1 expression was determined by IHC and strong PD-L1 positive was defined as a PD-L1 tumor proportion score ≥50%. OS was defined as the time from the first day of study treatment to death due to any cause. OS was analyzed by the Kaplan-Meier method for censored data and reported in months. Participant data were censored at last assessment.
Time Frame: Up to 76.9 months
Population: All participants who received at least one dose of study treatment with a tumor proportion score ≥50%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab
Number analyzed (Participants) | 44
Months | 6.9 [4.0 to 11.8]

ADVERSE EVENTS:
Time Frame: First Course: Up to 76.9 months Second Course: Up to 53.3 months First and second course dosing occurred concurrently
Description: All-cause mortality (ACM)=all allocated participants; AEs=all participants who received ≥1 dose of study treatment. Per protocol, disease progression was not considered an AE unless related to treatment. Medical Dictionary for Regulatory Activities (MedDRA) terms neoplasm progression, malignant neoplasm progression, and disease progression not related to treatment were excluded. Per protocol, collection of AEs and ACM were planned for both first and second courses.
Groups:
- Pembrolizumab Second Course: Participants who met the criteria for re-treatment received pembrolizumab 200 mg by IV infusion on Day 1 of each 3-week cycle for up to 1 year of treatment.
Arm/Group | Pembrolizumab | Pembrolizumab Second Course
All-Cause Mortality (participants affected / at risk) | 153/172 | 2/3
Serious Adverse Events (participants affected / at risk) | 87/171 | 1/3
Other Adverse Events (participants affected / at risk) | 158/171 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=171) | Pembrolizumab Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Swelling face (General disorders) | 2 (2) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 15 (18) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Cranial nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 0 (0)
Device dislocation (Product Issues) | 2 (2) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab (N=171) | Pembrolizumab Second Course (N=3)
Anaemia (Blood and lymphatic system disorders) | 32 (35) | 0 (0)
Hypothyroidism (Endocrine disorders) | 32 (34) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (13) | 0 (0)
Constipation (Gastrointestinal disorders) | 42 (46) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 24 (38) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 12 (12) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 23 (24) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 34 (37) | 0 (0)
Vomiting (Gastrointestinal disorders) | 15 (15) | 0 (0)
Fatigue (General disorders) | 67 (71) | 0 (0)
Oedema peripheral (General disorders) | 11 (13) | 0 (0)
Pyrexia (General disorders) | 10 (11) | 0 (0)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 12 (15) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 9 (10) | 0 (0)
Stoma site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 11 (13) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 19 (20) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 9 (9) | 1 (1)
Lymphocyte count decreased (Investigations) | 10 (10) | 0 (0)
Weight decreased (Investigations) | 33 (33) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 30 (36) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 16 (20) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 13 (15) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (23) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 (16) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 11 (13) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (16) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 (17) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 29 (41) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 (33) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (13) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 13 (14) | 0 (0)
Dizziness (Nervous system disorders) | 18 (21) | 0 (0)
Headache (Nervous system disorders) | 20 (20) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 9 (9) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 1 (1)
Insomnia (Psychiatric disorders) | 18 (19) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (39) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 (26) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 17 (20) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (7) | 1 (1)
Hypertension (Vascular disorders) | 11 (17) | 0 (0)
Hypotension (Vascular disorders) | 16 (17) | 0 (0)
Lymphoedema (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT02255097/Prot_SAP_000.pdf